CLINICAL TRIAL: NCT06037811
Title: Early Adalimumab Induction for Treatment of Steroid Dependent Immune Checkpoint Inhibitor Associated Inflammatory Arthritis: a Pragmatic Randomized Clinical Trial
Brief Title: Early Adalimumab Induction for Immune Checkpoint Inhibitor Associated Inflammatory Arthritis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tom Appleton (Other)
Collaborators: Canadian Research Group in Immuno-Oncology (Unknown); Western University (Other)
Responsible Party: Sponsor-Investigator, Tom Appleton, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CanRIO ADA2023
Record Dates: First submitted 2023-08-31; First posted 2023-09-14 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-03

CONDITIONS: Inflammatory Arthritis; Immune-related Adverse Event
Keywords: Immune Checkpoint Inhibitor; Adalimumab; TNF-alpha inhibitor
MeSH Terms: conditions — Arthritis | interventions — Adalimumab; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care group (Active Comparator): Prednisone 10 mg daily for 2 weeks, then taper by 2.5 mg every 2 weeks until stopped.
  Interventions: Drug: Prednisone
- Adalimumab group (Active Comparator): Adalimumab 40 mg subcutaneous every 2 weeks for 6 doses (12 weeks)
  + Prednisone 10 mg daily for 2 weeks, tapering by 2.5 mg every 2 weeks until stopped.
  Interventions: Drug: Adalimumab; Drug: Prednisone

INTERVENTIONS:
Drug: Adalimumab — Participants will be randomized 1:1 (non-blinded) to receive either adalimumab (40 mg subcutaneous every 2 weeks for 12 weeks) and prednisone vs prednisone alone. Addition of methotrexate (MTX) and/or hydroxychloroquine (HCQ) is permitted, as needed, at the discretion of the treating rheumatologist. No additional conventional synthetic, targeted synthetic or biologic DMARDs are permitted during the trial.
  Arms: Adalimumab group
Drug: Prednisone — Prednisone as per standard of care.

SUMMARY:
This study will examine the effectiveness of administering adalimumab as a treatment for patients in the early stages of steroid-dependent immune checkpoint Inhibitor associated inflammatory arthritis (ir-IA). Adalimumab (ADA) is a TNF inhibitor (TNFi) that is well established as a standard of care treatment for numerous types of inflammatory arthritis. It is hoped that adalimumab at the early stages of the ir-IA will reduce the symptoms and therefore reduce the need for steroids. This study is a pragmatic randomized clinical trial. Patients will be randomized 1:1 to each treatment group. To evaluate the steroid sparing effect of early induction six doses of Adalimumab will be administered to patients in the study treatment arm as compared to the usual standard of care of a predefined corticosteroid regimen and taper at 12 weeks administered in the control group.

ELIGIBILITY:
Inclusion Criteria:

* • Patients are deemed eligible for study participation if they meet all the following:

  * Adult patients (age 18 or older)
  * New (within the last 6 months prior to enrollment) inflammatory arthritis defined by any of the following at the time of screening (either on physical exam or by ultrasound) by a certified rheumatologist:
* 1 or more swollen joints OR
* 1 or more tenosynovitis OR
* 1 or more enthesitis

  * Arthritis onset with taking ICI therapy OR within 4 weeks of stopping ICI therapy including CTLA-4, PD-1, and PDL-1 inhibitors
  * Initiation of ICI therapy must predate the onset of inflammatory arthritis
  * Arthritis either does not respond completely to prednisone doses of 10mg (equivalent) OR recurs with prednisone taper below 10mg daily.
  * Negative tuberculosis (TB) status within the past 12 months (TB skin test or quantiferon) for the patients in the adalimumab group. If not available, the status should be confirmed within 6 months of enrollment in the study (adalimumab group only)
  * Written informed consent provided by patient or power of attorney

Exclusion Criteria:

* Patients are excluded if they meet any of the following:
* Previous diagnosis of inflammatory arthritis or other rheumatic disease (prior to current acute episode)

  * Including but not limited to: rheumatoid arthritis, systemic lupus erythematosus, systemic sclerosis, Sjogren's syndrome, psoriatic arthritis, reactive arthritis, ankylosing spondylitis, systemic vasculitis, undifferentiated inflammatory arthritis, undifferentiated connective tissue disease
* Tenosynovitis, synovitis or enthesitis attributed to another cause, fracture or acute gout/CPPD flare.
* Presence of a contraindication to adalimumab therapy

  * Any of the following in the 7 days prior to initiation of adalimumab: positive tuberculin skin test (>5mm induration within 48 to 72 hours) or positive quantiferon, evidence of untreated active infection including fungal infection, opportunistic infection, hepatitis B/C, or HIV
  * Personal history of congestive heart failure
  * Personal or family history of demyelinating neurologic disease
* History of previous TNF inhibitor use
* Current use of other disease modifying agents including: Chloroquine, Sulfasalazine, Azathioprine, 6-MP, and Leflunomide
* Presence of a concomitant non-rheumatic irAE which required systemic immunosuppression within the past 3 months e.g. pneumonitis, hepatitis, colitis, scleritis, nephritis
* Require chronic steroid treatment for adrenal insufficiency or another medical reason other than ir-IA
* Pregnancy, breastfeeding or childbearing potential without practicing highly effective contraception.
* Inability to participate in follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
percentage of participants on prednisone | at 12 weeks
  Definition of success: Thirty percent fewer participants on prednisone in Group 2 vs Group 1.
Cumulative prednisone dose | at 12 weeks
  Definition of success: Thirty percent reduction in the cumulative dose of steroids in Group 2 compared to Group 1.

SECONDARY OUTCOMES:
percentage of participants on prednisone | 24 weeks
  Definition of success: Thirty percent difference between the two groups
Cumulative prednisone dose | 24 weeks
  Definition of success: Thirty percent difference between the two groups
percentage of dose reduction of prednisone | At 12 and 24 weeks
  Definition of success: Thirty percent difference between the two groups
percentage of participants with immune-related inflammatory arthritis in remission (based on opinion of investigator) | at 12 and 24 weeks
  Definition of success: Thirty percent difference between the two groups
percentage of participants with immune-related inflammatory arthritis resolution (based on opinion of investigator) | at 12 and 24 weeks
  Definition of success: Thirty percent difference between the two groups

OTHER OUTCOMES:
percentage of participants with persistent active synovitis/tenosynovitis (yes/no) | at 12 and 24 weeks
  Differences between treatment groups ≥20% will be considered significant
percentage of participants treated with methotrexate and/or hydroxychloroquine | at 12 and 24 weeks
  Differences between treatment groups ≥20% will be considered significant
MDGA (MD global assessment) of arthritis 0 to 10 | at weeks 12 and 24
  Differences between treatment groups ≥20% will be considered significant
Participant reported pain on a visual analog scale from 0 to 10. | at weeks 12 and 24
  Enhancement of quality of life due to ADA will be defined as 50% improvement in any of these readouts in ≥50% of participants at weeks 12 and 24 compared to Group 1.
PGA (patient global assessment) of arthritis 0-10 | at weeks 12 and 24
  Enhancement of quality of life due to ADA will be defined as 50% improvement in any of these readouts in ≥50% of participants at weeks 12 and 24 compared to Group 1.
FACIT-F (Functional Assessment of Chronic Illness Therapy-Fatigue Score) | at weeks 12 and 24
  Enhancement of quality of life due to ADA will be defined as 50% improvement in any of these readouts in ≥50% of participants at weeks 12 and 24 compared to Group 1.
EQ-5D (EuroQol 5 Dimension for evaluation of generic quality of life) | at weeks 12 and 24
  Enhancement of quality of life due to ADA will be defined as 50% improvement in any of these readouts in ≥50% of participants at weeks 12 and 24 compared to Group 1.
Cancer status vs baseline: overall survival (OS), progression free survival (PFS) | at 12 and 24 weeks
  Differences between treatment groups ≥20% will be considered significant
Number of participants who continue, hold or stop ICI therapy | at 12 and 24 weeks
  Differences between treatment groups ≥20% will be considered significant
Feasibility: Number of participating sites; Number of participants screened, consented, randomized, and followed-up at each participating site | at week 24
  Differences between treatment groups ≥20% will be considered significant
The rates of AEs, serious AEs (according to CTCAE), and clinical laboratory abnormalities | at 12 and 24 weeks
  ADA will be considered 'safe' if the frequency of moderate AEs in Group 2 does not exceed 50% (reported rate of moderate AE in RA is 41%)

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Health Care, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided